CLINICAL TRIAL: NCT00062829
Title: Young Driver Intervention Study: Preventing Motor Vehicle Crashes Among Young Drivers
Brief Title: Young Driver Intervention Study: Preventing Motor Vehicle Crashes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Denise Haynie, Staff Scientist, Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: N01HD83285; Z01HD001707-01 (NIH); N01-HD-8-3285
Record Dates: First submitted 2003-06-17; First posted 2003-06-18 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Accidents, Traffic; Health Behavior
Keywords: Teen driving; Adolescent risk behavior; Parenting; Checkpoints Program; Health Education
MeSH Terms: conditions — Health Behavior; Health Education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Teen Driving: Program for parents (Other): A behavioral intervention targeting driving risks unique to young drivers, including completing a behavioral contract, was administered to the intervention group. The control group received safety information appropriate for new drivers.
  Interventions: Behavioral: Teen Driving: Program for parents

INTERVENTIONS:
Behavioral: Teen Driving: Program for parents — A behavioral intervention targeting driving risks unique to young drivers, including completing a behavioral contract, was administered to the intervention group. The control group received safety information appropriate for new drivers.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a program designed to reduce teen crashes and risky driving by increasing parental monitoring and restriction of their adolescents' driving practices during the first year of licensed driving.

DETAILED DESCRIPTION:
Motor vehicle crashes are the major cause of death and disability among adolescents from 16 through 20 years of age. While adolescents between the ages of 16 and 19 years constitute only 5% of all licensed drivers, they are involved in 15% of the crashes in which they or other occupants are killed. In fact, 16-year-old drivers are more than 20 times as likely to have a crash as the general population of drivers and 17-year-olds are more than 6 times as likely. In addition, for each adolescent motor vehicle fatality, approximately 100 nonfatal injuries occur, making crashes the leading cause of disability due to head and spinal cord injuries in adolescents.

Parents can have a huge impact on adolescent behavior. However, the impact of parenting practices on adolescent driving behavior has not yet been examined. This study aims to determine the efficacy of an intervention designed to increase parents' involvement in, and parental restrictions on, their teens' early driving experiences in order to reduce the number of tickets and crashes among teen drivers. The intervention provides educational materials to parents and adolescents from the time the adolescent gets a learner's permit through the first 6 months of licensure. These persuasive communications are tailored to adolescents' level of driving experience. The intervention materials make explicit the increased risk associated with adolescent driving and methods for reducing risk through increased parental involvement in and restriction of driving.

Participants were recruited in the Connecticut Department of Motor Vehicle offices as adolescents applied for their learner's permits. Participants were randomized to either the intervention group or the control group. The control group received standard information about driving not related to the specific teen risks focused on in the intervention group materials. All participants completed interviews at study entry, licensure, 3 months after licensure, 6 months after licensure, and 12 months after licensure. Parents were asked about their expectations and parenting practices regarding their adolescents' driving behaviors. Adolescents were asked about their driving practices and their parents' rules and restrictions regarding driving. The driving records for each adolescent were obtained from the state motor vehicle administration and examined 18 months after licensure.

ELIGIBILITY:
Inclusion Criteria

* Lives with parent/guardian at least 50% of the time
* Obtains learner's driving permit
* Family members are able to complete interviews in English

Ages: 16 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3743 (Actual)
Dates: Start 1998-09; Primary Completion 2000-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Risky Driving | 12 months
  17 item assessment of engaging in risky driving behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Simons-Morton, EdD, MPH, Principal Investigator — Prevention Research Branch, Division of Epidemiology, Statistics and Prevention Research, NICHD

REFERENCES:
- [Background] Simons-Morton BG, Hartos JL. How well do parents manage young driver crash risks? J Safety Res. 2003 Jan;34(1):91-7. doi: 10.1016/s0022-4375(02)00085-3. PMID 12535911
- [Background] Simons-Morton BG, Hartos JL, Leaf WA. Promoting parental management of teen driving. Inj Prev. 2002 Sep;8 Suppl 2(Suppl 2):ii24-30; discussion ii30-1. doi: 10.1136/ip.8.suppl_2.ii24. PMID 12221027
- [Background] Simons-Morton BG. Reducing young driver crash risk. Inj Prev. 2002 Sep;8 Suppl 2(Suppl 2):ii1-2. doi: 10.1136/ip.8.suppl_2.ii1. No abstract available. PMID 12221023